CLINICAL TRIAL: NCT04218838
Title: A Prospective, Multi-Center, Bi-Phasic Randomized Design to Compare Outcomes of the CornerLoc™ SI Joint Stabilization System and Intra-Articular Sacroiliac Joint Steroid Injection in Patients With Refractory Sacroiliac Joint Dysfunction
Brief Title: Comparison of CornerLoc SI Joint Stabilization and Steroid Injections for Sacroiliac Joint Dysfunction
Acronym: COVI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment difficulties due to changes in control arm conventions
Sponsor: CornerLoc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: COVI-0001
Record Dates: First submitted 2019-12-30; First posted 2020-01-06 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Sacroiliac Joint Somatic Dysfunction

STUDY DESIGN:
Intervention Model Description: Within the initial phase, referred to as the Randomized Phase, the primary determination of efficacy and safety will be 6-months following the study procedure. The analysis will be based on the randomization assignment. In the second phase of the study, referred to as the Cross-over Phase, patients who fail to respond to the randomized treatment assignment will be permitted to receive the non-randomized treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- CornerLoc SI Joint Stabilization Group (Active Comparator): Patient will receive the CornerLoc minimally invasive SI Joint Stabilization procedure. This procedure will be performed in an outpatient surgery center under local sedation or general anesthesia, and normally takes around 45 minutes. During the procedure, the physician will make two small incisions in the patient's lower back to access the SI joint, and place four small cadaveric bone grafts into the SI joint to help stabilize the SI joint.
  Interventions: Device: CornerLoc SI Joint Stabilization Procedure
- SI Joint Steroid Injections Group (Active Comparator): Patient will receive an injection of steroid medication directly into their SI joint. The area around the SI joint will be numbed with an injection of local anesthetic and then ultrasound guidance will be used to guide the needle of steroid medication directly into the SI joint. This procedure will be performed in the physician's office or an outpatient surgery center, and normally takes around 30 minutes.
  Interventions: Drug: Intra-articular Sacroiliac Joint Steroid Injection

INTERVENTIONS:
Device: CornerLoc SI Joint Stabilization Procedure — CornerLoc minimally invasive SI Joint Stabilization System
  Arms: CornerLoc SI Joint Stabilization Group
Drug: Intra-articular Sacroiliac Joint Steroid Injection — Standard of Care - Steroid injection into the sacroiliac joint
  Arms: SI Joint Steroid Injections Group

SUMMARY:
This study has been designed to compare the safety and effectiveness of the CornerLoc™ SI Joint Stabilization System to intra-articular sacroiliac joint steroid injection in patients with refractory sacroiliac joint dysfunction.

DETAILED DESCRIPTION:
Randomized, multicenter, open-label, randomized design to compare CornerLoc Allograft-based Sacroiliac Joint Stabilization System to Intra-articular Sacroiliac Joint Steroid Injection. Within the initial phase, referred to as the Randomized Phase, the primary determination of efficacy and safety will be 6-months following the study procedure. The analysis will be based on the randomization assignment. In the second phase of the study, referred to as the Cross-over Phase, patients who fail to respond to the randomized treatment assignment will be permitted to receive the non-randomized treatment. The basis of the sample size and hypothesis testing for this clinical investigation will be based on the Randomization Phase.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following inclusion criteria by the end of the screening phase should be considered for admission to the study:

  * Subject must provide written informed consent prior to any clinical study-related procedure.
  * Subject is at least 18 years (or the minimum age required by local law to consent for participation in a clinical investigation) or older at the time of enrollment.
  * Subjects must meet criteria for sacroiliac joint dysfunction as determined below:
  * History of persistent pain in the distribution of the sacroiliac joint despite adequate trial of physical therapy.
  * NRS for pain ≥ 7 on a 0 -.10-point scale.
  * 3 of 5 provocative tests with positive findings on physical examination (SI distraction, thigh thrust, FABER, lateral compression, Gaenslen's maneuver).
  * Positive response (≥75% percent pain relief) to diagnostic sacroiliac joint injection on two occasions at least one week apart.
  * Baseline pain with 30-day history and PROMIS-29

Exclusion Criteria:

* Patient will not be entered into the study if they meet one of the following criteria:

  * Subject is unable to provide written informed consent
  * Subject is enrolled, or intends to participate, in a clinical drug and/or device study (investigational device, investigational drug, new indication for a device or drug, or additional testing beyond standard of care procedures) which could confound the results of this trial as determined by the investigator.
  * Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
  * Subject had prior surgical fusion implanted on same side
  * Subject is pregnant or nursing
  * Self-reported plan to bear children
  * BMI ≥ 40
  * DEXA < -2.5 (if available)
  * History of microfractures
  * History of compression fractures
  * History of diabetes, must have A1c <8
  * History of chronic steroid use
  * Chronic immunosuppression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of sacroiliac joint stabilization using the CornerLoc procedure in the treatment of sacroiliac joint pain by evaluating the efficacy responder rate versus an intra-articular steroid injection. | 6 months
  The efficacy responder rate is defined as the percentage of subjects who experience at least a 50% improvement in overall pain, as measured by the Numeric Rating Scale (NRS) for Pain, from Baseline to the 6-Month Visit. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Quality of life improvement from baseline to each follow-up visit. | 6 months
  PROMIS-29; Patient Reported Outcomes Measurement Information System (PROMIS) instruments contain a fixed number of items from seven PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. The seven domains cover the most relevant areas of self-reported health for the greatest majority of people with chronic illness.
  The PROMIS-29, a generic health-related quality of life survey, assesses each of the 7 PROMIS domains with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity.
Clinical improvement based on pain from baseline to each follow-up visit. | 6 months
  Numeric Rating Scale for Pain: The Numeric Rating Scale for Pain is a measure in which individuals rate their pain on an eleven point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). The patient will be asked to point to the number on the Numeric Rating Scale that best represents intensity of pain.
Clinical improvement of low back pain from baseline to each follow-up visit. | 6 months
  Oswestry Disability Index (ODI): The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is a tool for evaluators used to measure a patient's permanent functional disability. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability. The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). A higher score on the ODI indicates a more severe disability caused by lower back pain.
Clinical improvement in balance and risk for falls from baseline to each follow-up visit. | 6 months
  Timed Up and Go" (TUG) Test: This test measures the time for a subject to get up from a chair walk 3 meters, turn around and return to the chair and sit. Time is measured in minutes and seconds. An average of two tests is used. The shorter average time indicates clinical improvement.
Clinical improvement from baseline to each follow-up visit. | 6 months
  Zurich Claudication Questionnaire (ZCQps); The Zurich Claudication Questionnaire quantifies severity of symptoms, physical function characteristics, and patient's satisfaction after treatment. The scale relates to symptoms over the past month. There are 12 questions for all patients, and a further 6 questions to measure treatment outcome. Decreasing scores indicates clinical improvement
Clinical improvement based on use of medications from baseline to each follow-up visit. | 6 months
  Medication Use: All medications that are used prior to and during their participation in this study will be documented and monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fishman, MD, Principal Investigator — Center for Interventional Pain & Spine
Locations (1):
- Center for Interventional Pain and Spine, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No